CLINICAL TRIAL: NCT01198548
Title: A Phase II Clinical Trial of High Dose Vitamin D3 Supplementation in Combination With FOLFOX + Bevacizumab in the 1st Line Treatment of Metastatic Colorectal Cancer
Brief Title: High-Dose Cholecalciferol in Treating Patients Receiving Combination Chemotherapy and Bevacizumab as First-Line Therapy For Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 176910; NCI-2010-01783 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2010-09-08; First posted 2010-09-10 (Estimated); Results first posted 2014-07-21 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-06

CONDITIONS: Stage IV Colon Cancer; Stage IV Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Leucovorin; Bevacizumab; Cholecalciferol; Fluorouracil; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (FOLXFOX, bevacizumab, cholecalciferol) (Experimental): Patients receive high-dose cholecalciferol once daily. Patients also receive bevacizumab IV over 10 minutes, leucovorin calcium IV over 2 hours, oxaliplatin* IV over 2 hours, and fluorouracil IV continuously over 46 hours once a week. Courses repeat every 2 weeks in the absence of disease progression or unacceptable toxicity. NOTE: *Treatment with oxaliplatin is discontinued after course 8
  Interventions: Drug: leucovorin calcium; Biological: bevacizumab; Dietary Supplement: cholecalciferol; Drug: fluorouracil; Drug: oxaliplatin; Other: pharmacological study

INTERVENTIONS:
Drug: leucovorin calcium — Given IV
  Other Names: CF; CFR; LV
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Dietary Supplement: cholecalciferol — Given PO
  Other Names: Calciol; Vitamin D3
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase II trial is studying how well giving high-dose cholecalciferol works in treating patients receiving combination chemotherapy and bevacizumab as first-line therapy for metastatic colorectal cancer. Cholecalciferol during treatment may delay the development of colorectal cancer. Drugs used in chemotherapy, such as leucovorin calcium, fluorouracil, and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving cholecalciferol together with combination chemotherapy and monoclonal antibody therapy may be an effective treatment for colorectal cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the relative rate of metastatic colorectal cancer patients who achieve 25-D3 levels >= 40 ng/ml at 8 weeks, 16 weeks, 24 weeks, and 32 weeks from starting FOLFOX (leucovorin calcium, fluorouracil, and oxaliplatin) + bevacizumab + high dose vitamin D3 supplementation (cholecalciferol).

II. To estimate the median progression-free survival (PFS) of metastatic colorectal cancer patients receiving first-line FOLFOX + bevacizumab + high dose vitamin D3 supplementation.

SECONDARY OBJECTIVES:

I. To estimate the response rate (RR) and the median overall survival (OS) of metastatic colorectal cancer patients receiving first-line FOLFOX + bevacizumab + high dose vitamin D3 supplementation.

II. To describe the safety of this combination by capturing all treatment-related toxicity as per National Cancer Institute-Common Terminology Criteria (NCI-CTC) version 4 guidelines.

OUTLINE:

Patients receive high-dose cholecalciferol orally (PO) once daily. Patients also receive bevacizumab intravenously (IV) over 10 minutes, leucovorin calcium IV over 2 hours, oxaliplatin* IV over 2 hours, and fluorouracil IV continuously over 46 hours once a week. Courses repeat every 2 weeks in the absence of disease progression or unacceptable toxicity.

NOTE: *Treatment with oxaliplatin is discontinued after course 8.

After completion of study treatment, patients are followed up at day 30 and then 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients should have untreated metastatic colorectal cancer; prior adjuvant chemotherapy is allowed as long as the development of metastatic disease occurred more than 6 months from completion of adjuvant treatment
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
* Platelets >= 100,000/mm^3
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Hemoglobin > 9 gm/dl
* Calculated creatinine clearance > 40 ml/min according to the Cockcroft-Gault formula OR per 24 hour urine collection
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 2.5 x institutional upper normal level if no liver metastases and < 5 x upper limit of normal (ULN) in the setting of liver metastases
* Total bilirubin =< 1.5 x institutional upper normal level
* Albumin >= 2.5 g/dl
* Urine protein:creatinine (UPC) ratio < 1; in the event UPC is > 1, the patient will require a 24-hr urine protein and will be eligible if 24-hr urine collection has < 1,000 mg protein
* Patients of child-hearing potential must agree to use acceptable contraceptive methods (e.g., double harrier) during treatment
* Patient or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board-approved written informed consent form prior to receiving any study-related procedure
* Presence of measurable disease defined as a lesion >= 1 cm by computed tomography (CT); all sites of disease should be evaluated =< 3 weeks before treatment initiation
* Baseline 25-D3 level of < 40 ng/ml

Exclusion Criteria:

* Patients may not be receiving any other investigational agents that are not included in this study
* Patients with known brain metastases
* History of other invasive cancers with the exception of the following: a. Curatively resected or treated non-melanoma skin cancer; b. Curatively treated cervical carcinoma in situ; c. Other primary solid tumors treated curatively and no treatment administered >= 2 years before enrollment, and in the investigator opinion, it is unlikely that there will be a recurrence =< 1 year post enrollment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to oxaliplatin, 5-FU, leucovorin, bevacizumab, and vitamin D3 and other agents used in study
* History of clinically significant bleeding within 6 months of enrollment
* Clinically significant cardiovascular disease within 12 months prior to enrollment, including myocardial infarction, unstable angina, grade 2 or greater peripheral vascular disease, cerebrovascular accident, transient ischemic attack, congestive heart failure or arrhythmias not controlled by outpatient medication, percutaneous transluminal coronary angioplasty/stent
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated on this study
* Major surgery within 28 days prior to enrollment or still recovering from prior surgery
* Known dihydropyrimidine dehydrogenase (DpD) deficiency
* History or evidence upon physical examination of central nervous system (CNS) disease (e.g., primary brain tumor, seizures not controlled with standard medical therapy, any brain metastases, or history of stroke)
* Serious, nonhealing wound, ulcer, or bone fracture
* Uncontrolled hypertension (systolic blood pressure > 150 mmHg or diastolic blood pressure > 95 mmHg despite medications)
* History of arterial thrombosis within the last 12 months
* History of visceral arterial ischemia
* Subjects unwilling or unable to comply with study requirements
* Any condition that in the Investigator's opinion deems the patient an unsuitable candidate to receive study drug
* Received an investigational agent within 30 clays prior to enrollment
* Treatment with vitamin D replacement with doses exceeding an average of 1000 IU/day (vitamin D3) within 60 days prior to enrollment

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-08; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wen Wee Ma, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (FOLXFOX, Bevacizumab, Cholecalciferol)
Started | 10
Completed | 0
Not Completed | 10
Not completed — Disease Progression | 9
Not completed — Administrative Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (FOLXFOX, Bevacizumab, Cholecalciferol)
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (8.43)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Median PFS
Description: The estimated distributions of PFS will be obtained using the product-limit based Kaplan-Meier method. The corresponding 95% confidence intervals for the estimated probability will be computed using the method proposed in Clopper and Pearson.
Time Frame: Up to 12 months
Population: Due to the study's early termination and inadequate number of patients, no patients were analyzed.
Arm/Group | Treatment (FOLXFOX, Bevacizumab, Cholecalciferol)
Number analyzed (Participants) | 0

2. Primary Outcome: Rate of Sufficient Cholecalciferol
Time Frame: By week 16
Population: Due to the study's early termination and inadequate number of patients, no patients were analyzed.
Arm/Group | Treatment (FOLXFOX, Bevacizumab, Cholecalciferol)
Number analyzed (Participants) | 0

3. Secondary Outcome: RR of Patients Receiving Study Treatment
Time Frame: Up to 3 years
Population: Trial terminated early. Too few patients to analyze.
Arm/Group | Treatment (FOLXFOX, Bevacizumab, Cholecalciferol)
Number analyzed (Participants) | 0

4. Secondary Outcome: Toxicity Rates as Assessed by NCI CTCAE Version 4
Time Frame: Up to 30 days post-treatment
Population: Due to the study's early termination and inadequate number of patients, no patients were analyzed.
Arm/Group | Treatment (FOLXFOX, Bevacizumab, Cholecalciferol)
Number analyzed (Participants) | 0

5. Secondary Outcome: OS of Patients Receiving Study Treatment
Description: The estimated distribution of OS will be obtained using the product-limit based Kaplan-Meier method.
Time Frame: Up to 3 years
Population: Due to the study's early termination and inadequate number of patients, no patients were analyzed.
Arm/Group | Treatment (FOLXFOX, Bevacizumab, Cholecalciferol)
Number analyzed (Participants) | 0

6. Secondary Outcome: PFS of Patients Receiving Study Treatment
Description: The estimated distributions of PFS will be obtained using the product-limit based Kaplan-Meier method.
  3 Year Survival Rate
Time Frame: Defined as the time from the start of the study treatment until the date of progression or death from any cause, whichever comes first, assessed up to 3 years
Population: Due to the study's early termination and inadequate number of patients, no patients were analyzed.
Arm/Group | Treatment (FOLXFOX, Bevacizumab, Cholecalciferol)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Treatment (FOLXFOX, Bevacizumab, Cholecalciferol)
Serious Adverse Events (participants affected / at risk) | 4/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (FOLXFOX, Bevacizumab, Cholecalciferol) (N=10)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (12)
Abdominal pain (Gastrointestinal disorders) | 1 (6)
Intestinal obstruction (Gastrointestinal disorders) | 1 (6)
Nausea (Gastrointestinal disorders) | 1 (6)
Pancreatitis (Gastrointestinal disorders) | 1 (10)
Pyrexia (General disorders) | 1 (6)
Hypersensitivity (Immune system disorders) | 1 (6)
Infection (Infections and infestations) | 1 (6)
Urinary tract infection (Infections and infestations) | 1 (6)
Wound infection (Infections and infestations) | 1 (12)
Renal failure acute (Renal and urinary disorders) | 1 (12)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (5)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (FOLXFOX, Bevacizumab, Cholecalciferol) (N=10)
Anaemia (Blood and lymphatic system disorders) | 2 (17)
Leukopenia (Blood and lymphatic system disorders) | 3 (42)
Lymphopenia (Blood and lymphatic system disorders) | 1 (6)
Neutropenia (Blood and lymphatic system disorders) | 6 (48)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (6)
Abdominal pain (Gastrointestinal disorders) | 1 (5)
Cheilitis (Gastrointestinal disorders) | 1 (6)
Constipation (Gastrointestinal disorders) | 1 (6)
Diarrhoea (Gastrointestinal disorders) | 5 (27)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (12)
Nausea (Gastrointestinal disorders) | 2 (16)
Oesophageal pain (Gastrointestinal disorders) | 1 (5)
Oral pain (Gastrointestinal disorders) | 1 (5)
Proctalgia (Gastrointestinal disorders) | 1 (10)
Stomatitis (Gastrointestinal disorders) | 1 (6)
Vomiting (Gastrointestinal disorders) | 2 (22)
Fatigue (General disorders) | 2 (14)
Mucosal inflammation (General disorders) | 1 (6)
Pain (General disorders) | 1 (6)
Pyrexia (General disorders) | 1 (5)
Skin infection (Infections and infestations) | 1 (5)
Tooth abscess (Infections and infestations) | 1 (5)
Limb injury (Injury, poisoning and procedural complications) | 1 (4)
Blood alkaline phosphatase increased (Investigations) | 3 (20)
Blood amylase increased (Investigations) | 1 (5)
Haemoglobin (Investigations) | 1 (5)
Lipase increased (Investigations) | 1 (5)
Weight decreased (Investigations) | 1 (6)
Anorexia (Metabolism and nutrition disorders) | 1 (6)
Hyperalbuminaemia (Metabolism and nutrition disorders) | 1 (6)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (16)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (11)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (6)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (5)
Dysgeusia (Nervous system disorders) | 1 (6)
Headache (Nervous system disorders) | 2 (12)
Neuropathy peripheral (Nervous system disorders) | 1 (5)
Proteinuria (Renal and urinary disorders) | 1 (5)
Genital pruritus female (Reproductive system and breast disorders) | 1 (5)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (6)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (6)
Hypertension (Vascular disorders) | 3 (25)
Hypotension (Vascular disorders) | 1 (5)

LIMITATIONS AND CAVEATS:
Due to the study's early termination and inadequate number of patients, no patients were analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes